CLINICAL TRIAL: NCT03984721
Title: Amyloidosis Typing Using Mass Spectrometry-based Proteomics: a New Accurate Tool for Difficult Typing
Acronym: TYPAMYL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/16/8768
Record Dates: First submitted 2019-06-05; First posted 2019-06-13 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Amyloidosis
Keywords: Mass spectrometry based proteomic analysis; NanoLC-MS/MS; Amyloidosis typing
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Intervention Model Description: Inclusion of 40 patients identified by the Department of Anatomy and pathological cytology at the University of Toulouse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amylose typing (Experimental): Amyloidosis typing by nanoLC-MS/MS in patients diagnosed with Amyloidosis but unable to be typed
  Interventions: Diagnostic Test: Amyloidosis typing using mass spectrometry-based proteomics

INTERVENTIONS:
Diagnostic Test: Amyloidosis typing using mass spectrometry-based proteomics — Amyloidosis typing using nanoLC-MS/MS method

SUMMARY:
The main objective is to establish that a new technique of amyloidosis typing by Proteomics (based on nanoLC-MS/MS mass spectrometry) allows typing in > 90% of observations in patients whose Amyloidosis is reported to have failed typing (impossible typing, uncertain or inconsistent) with the traditional anatomopathological approach, and this in a cohort of 40 patients identified consecutively in the Department of pathological anatomy and cytology of the University Hospital of Toulouse and included prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Amyloidosis by Red Congo staining and birefringence in polarized light on tissue sampling
* Immunolabeling Amyloidosis typing

  1. impossible (no frozen sample available)
  2. or inconclusive (doubtful)
  3. or inconsistent with clinical, biological, genetic and iconographic data
* Signature of the informed consent form

Exclusion Criteria:

* Insufficient tissue material to perform the new technique
* Person placed under judicial protection
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Amyloidosis typing | Day 0
  Amyloidosis typing rate with the new technique

SECONDARY OUTCOMES:
Time to return the result | Day 0
  Time to return the result with the new technique (time in days)
Concordance | Day 0
  Agreement between the proteomic conclusion and the clinical judgement (binary answer : yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique CHAUVEAU, Principal Investigator — CHU Rangueil
Locations (1):
- University hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vrana JA, Gamez JD, Madden BJ, Theis JD, Bergen HR 3rd, Dogan A. Classification of amyloidosis by laser microdissection and mass spectrometry-based proteomic analysis in clinical biopsy specimens. Blood. 2009 Dec 3;114(24):4957-9. doi: 10.1182/blood-2009-07-230722. Epub 2009 Oct 1. PMID 19797517
- [Background] Theis JD, Dasari S, Vrana JA, Kurtin PJ, Dogan A. Shotgun-proteomics-based clinical testing for diagnosis and classification of amyloidosis. J Mass Spectrom. 2013 Oct;48(10):1067-77. doi: 10.1002/jms.3264. PMID 24130009